CLINICAL TRIAL: NCT06503952
Title: Impact of Uterine Immune Profiling and Personalized Treatments on Subsequent Live Birth in Patients Receiving a Single Blastocyst: a Matched Controlled Study
Brief Title: Impact of Uterine Immune Profiling and Personalized Treatments in Patients Receiving a Single Blastocyst: a Matched Controlled Study
Acronym: UTIMPROSET
Status: Not yet recruiting | Type: Observational
Sponsor: Matricelab Innove (Other)
Responsible Party: Principal Investigator, Dr Nathalie Lédée, MD, PhD, Matricelab Innove
Other Study IDs: MatriceLab Innove
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Infertility; Success Rate of Assisted Reproductive Therapy; Single Embryo Transfer; Pregnancy Outcomes; Immunological Tolerance; Immune System
Keywords: infertility; success rate of assisted reproductibve therapy; Single embryo transfer; uterine immune profiling; personalized care; Live birth rate
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- case group: Case group: All the patients who would have benefitted (with informed consent) of a uterine immune profile and a fresh Day-5 SET or a day-5 or-6 SET between January 2020 and march 2024 would be enrolled
- control group: Pair-matched group: Group without uterine immune profile before the SET Matching criteria will be maternal age (+/-1year) and, number of previous egg retrievals (including the ones without any transfer) and, number of previous ETs and technique used (IVF, ICSI, frozen embryo transfer) and degree of expansion of blastocoel (B1-B2/B3-B4/B5-B6) to reflect the quality of the embryo transferred

SUMMARY:
A recent randomised controlled trial and previous large cohort studies have shown that the uterine immune environment is a crucial element in improving the performance of Assisted Reproductive therapy (ART). As previous studies mixed Day-3, Day-5, single or doble embryo transfer, the clear influence of the endometrial environment on the embryo itself and its type of transfer (fresh or freeze thawed) need further investigation.

To complement previous studies, the present matched- pair study aims to select the population who exclusively received a single Day-5 embryo transfer (SET) and benefitted of a uterine immune profiling between 1 January 2020 and 30 June 2023 before the SET Day-5.

This population will be matched to a population. who did not have uterine immune profiling in the nine months prior to the single Day 5 embryo transfer between 2018 and 2023.

The matching criteria are the maternal age (+/-1 year), the past history of ART (same number of previous oocytes pick-up, same number of previous embryo transfer) and the same type of transfer (IVF, ICSI, frozen transfer) and the same category of expansion of the blastocoel (B1-B2/ B3-B4/ B5-B6).

The primary end-point is the live birth rate (LBR) following the Day 5 SET in the population who benefited from pre-SET immune profiling versus the LBR following the Day 5 SET in the pair- matched population who did not benefit from pre-SET uterine immune profiling Secondary end point are the clinical pregnancy rate and miscarriage rate per SET in the two paired populations

DETAILED DESCRIPTION:
The PRECONCEPTIO software will be used to extract all the uterine immune profiles carried out between January 2020 and June 2023 for patients attending the two reproductive centres, Bluets and Diaconnesse.

In parallel, data will be extracted from the MEDIFIRST software selecting all patients who benefited from a single day 5 embryo transfer between January 2018 and March 2024.

The case group represents the selection of patients who had both uterine immune profiling prior to ET and Day 5 single embryo transfer within the nine months following uterine immune profiling.

Each patient in the treated group is matched to patients who had a single Day 5 ET without immune profiling in the nine months prior to ET.

Matching criteria will be maternal age (+/-1year) and, number of previous egg retrievals (including the ones without any transfer) and, number of previous ETs and technique used (IVF, ICSI, frozen embryo transfer) and degree of expansion of blastocoel (B1-B2/B3-B4/B5-B6) to reflect the quality of the embryo transferred The primary end-point is the live birth rate (LBR) following the Day 5 SET in the population who benefited from pre-SET immune profiling versus the LBR following the Day 5 SET in the pair- matched population who did not benefit from pre-SET uterine immune profiling Secondary end point are the clinical pregnancy rate and miscarriage rate per SET in the two paired populations

Impact of the uterine immune profiling on the live birth rate

* In function of the type of embryo transfer (fresh or freezed thawed)
* In function of the quality of the blastocyst transferred
* In function of the range of embryo transfer

ELIGIBILITY:
For case: Uterine immune profiling followed by a Day-5 fresh SET or day-5 or Day-6 freeze-thawed SET within the nine months following the uterine immune profiling between January 2020 and June 2023.

Will be excluded patients with no SET day-5, with uterine immune profiling more than nine months before, or with no matching pair For control: Blastocyst SET without uterine immune profiling within the year prior the embryo transfer matched to the case group between January 2018 on June 2023

* maternal age (+/-1 year) and
* the past history of ART (same number of previous oocytes pick-up, same number of previous embryo transfer) and
* the same type of transfer (IVF, ICSI, frozen transfer) and
* the same category of expansion of the blastocoel (B1-B2/ B3-B4/ B5-B6).

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female involved in IVF
Study Population: Patients with a single embryo transfer at Day-5 case group: With an immune profile within the nine month before ET Control group: without immune profiling performed
Sampling Method: Non-Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2025-01-15 (Estimated); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Live birth rate following the single Day-5 embryo transfer (ET) | 9 months after the ET
  Live birth rate following the Day-5 ET between the case and control groups

SECONDARY OUTCOMES:
Implantation rate following the Day-5 ET | one month after ET
  Implantation rate following the Day-5 ET between the case and control groups
Clinical pregnancy rate after the Day-5 ET | two weeks after ET
  Clinical pregnancy rate after the Day-5 ET between the case and control groups
Ongoing PR after the day-5 ET | 12 weeks after ET
  Ongoing PR after the day-5 ET between the case and control groups
Miscarriage rate after ET | 20 weeks after the ET
  Miscarriage rate after the Blastocyst SET in the case and the pair-matched group

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hopital des Bluets- centre d'assistance medicale à la procreation, Paris, Ile de
  - Hopital des diaconnesse- Centre d'assistance medicale a la procreation, Paris, Île-de-France Region

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: review on uterine immune profiling — https://pubmed.ncbi.nlm.nih.gov/37511080/
- See also: cohort study on uterine immune profiling — https://pubmed.ncbi.nlm.nih.gov/33841443/